CLINICAL TRIAL: NCT00053092
Title: National Mantle Cell Lymphoma Trial - Phase II Randomized Study of Fludarabine/Cyclophosphamide Combination With or Without Rituximab in Patients With Untreated Mantle Cell Lymphoma
Brief Title: Combination Chemotherapy With or Without Rituximab in Treating Patients With Mantle Cell Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Australasian Leukaemia and Lymphoma Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000269136; NCRI-LY05; ALLG-LY05; EU-20230; NCRILG-LY05
Record Dates: First submitted 2003-01-27; First posted 2003-01-28 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2007-06

CONDITIONS: Lymphoma
Keywords: contiguous stage II mantle cell lymphoma; noncontiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; stage III mantle cell lymphoma; stage IV mantle cell lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Mantle-Cell | interventions — Rituximab; Cyclophosphamide; fludarabine phosphate

INTERVENTIONS:
Biological: rituximab
Drug: cyclophosphamide
Drug: fludarabine phosphate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies such as rituximab can locate cancer cells and either kill them or deliver cancer-killing substances to them without harming normal cells. It is not yet known if combination chemotherapy is more effective with or without rituximab in treating mantle cell lymphoma.

PURPOSE: Randomized phase II trial to compare the effectiveness of fludarabine and cyclophosphamide combined with rituximab to that of fludarabine and cyclophosphamide alone in treating patients who have mantle cell lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the response rates in patients with previously untreated mantle cell lymphoma treated with fludarabine and cyclophosphamide with or without rituximab.
* Compare the time to disease progression in patients treated with these regimens.
* Compare the toxicity of these regimens, in terms of adverse event profile, in these patients.
* Compare the overall survival of patients treated with these regimens.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to 1 of 2 treatment arms:

* Arm I: Patients receive fludarabine IV* and cyclophosphamide IV* on days 1-3.
* Arm II: Patients receive rituximab IV on day 1 and fludarabine IV* and cyclophosphamide IV* on days 2-4.

NOTE: *In both arms, fludarabine and cyclophosphamide may be administered orally instead of IV.

Treatment repeats every 28 days for 2-8 courses in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 56-82 patients (28-41 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed previously untreated mantle cell lymphoma requiring therapy

  * Any stage

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* Not specified

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 2.5 times upper limit of normal (ULN)^*
* Alkaline phosphatase no greater than 2.5 times ULN^*
* Hepatitis B and hepatitis C negative NOTE: *Unless related to lymphoma

Renal

* Creatinine no greater than 2.5 times ULN^* NOTE: *Unless related to lymphoma

Other

* No other malignancy within the past 5 years except non-melanoma skin cancer or curatively resected carcinoma in situ of the cervix
* No prior psychological illness or condition that would preclude study compliance
* No known hypersensitivity to murine proteins
* No concurrent uncontrolled medical conditions
* No other illness that would severely limit life expectancy
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 6 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* No prior chemotherapy

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2002-10; Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Response rate
Time to disease progression
Toxicity
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Simon Rule, MD, Study Chair — Derriford Hospital; John Seymour, MD, Study Chair — Peter MacCallum Cancer Centre, Australia
Locations (2):
- Peter MacCallum Cancer Centre, East Melbourne, Victoria, Australia
- Derriford Hospital, Plymouth, England, United Kingdom

REFERENCES:
- [Result] Eve HE, Linch D, Qian W, Ross M, Seymour JF, Smith P, Stevens L, Rule SA. Toxicity of fludarabine and cyclophosphamide with or without rituximab as initial therapy for patients with previously untreated mantle cell lymphoma: results of a randomised phase II study. Leuk Lymphoma. 2009 Feb;50(2):211-5. doi: 10.1080/10428190802688509. PMID 19197729